CLINICAL TRIAL: NCT02750475
Title: Human Phototoxicity Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18851
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): All subjects are patched.
  Interventions: Drug: Sunscreen Sport Lotion (BAY987516); Other: Untreated Skin

INTERVENTIONS:
Drug: Sunscreen Sport Lotion (BAY987516) — 50 μl/cm*2 or 0.05 gm/cm*2 of each test product is applied to duplicate skin sites (approximately 2 x 2 cm each). After the test articles have dried for 5 to 15 min, the sites are covered by the appropriate patch.24 hours later, the set of patches covering the product are removed. Three (3) μl/ cm2 or 0.003 gm/cm*2 of the test product is reapplied to the test site, air dried for 5 to 15 minutes for volatilization and then the test site is exposed to UVA radiation.(Formulation number - RB# Y65-110)
Other: Untreated Skin — This site is patched without treatment as irradiated control

SUMMARY:
To determine the phototoxic potential of a topically applied article in human subjects

ELIGIBILITY:
Inclusion Criteria:

* be male or female between the ages of 18 and 60 inclusive;
* be lightly pigmented (Fitzpatrick Skin Type I, II, III);
* have read and signed the written Informed Consent Form and have completed a Health Insurance Portability and Accountability Act (HIPAA) Authorization Form in conformance with 45CFR Parts 160 and 164;
* be in general good health as determined by the subject's medical history and in the discretion of the investigator;

Exclusion Criteria:

* have a visible sunburn;
* have a history of sun hypersensitivity/photosensitivity or photosensitive dermatoses;
* must not have a known sensitivity or allergy against any of the active and non-active ingredients of the test product;
* have a history of allergies or sensitivities to cosmetics, toiletries or any dermatological products;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2016-05-06 (Actual)

PRIMARY OUTCOMES:
Intensity of skin reactions will be evaluated using the 5 point grading scale | Up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Piscataway, New Jersey, United States